CLINICAL TRIAL: NCT06240338
Title: Acute Pancreatitis : Comparison of Various Scores in Predicting Severity and Outcome
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ali Bakr Ahmed, Principal Investigator of tropical medicine, Sohag University
Other Study IDs: Soh-Med-23-12-05MD
Record Dates: First submitted 2024-01-02; First posted 2024-02-05 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: laboratory investigation and Imaging — laboratory parameters (white blood cell count,neutrophil count, lymphocyte count, hemoglobin level, platelet level, red cell distribution width (RDW) level, hematocrit (HCT), renal function, hepatic function, electrolytes, arterial blood gas, HOMA-IR) will be assessed and imaging: Abdominal ultrasonography, Abdominal CT or MRI if needed

SUMMARY:
The study will make a comparison between Various severity scoring systems that has been designed to assess the severity and predict prognosis in acute pancreatitis

DETAILED DESCRIPTION:
the study will evaluate the relationship between homeostatic model assessment of insulin resistance , bedside index of severity score and the harmless acute pancreatitis score and prognosis of acute pancreatitis ,will compare of these scores in predicting severity of acute pancreatitis and will compare of these scores in predicting outcome of acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with 18 years or above and met criteria for diagnosis of acute pancreatitis will be eligible for the study.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * age <18 years old,
  * patients with metastatic tumor
  * late stage of liver cirrhosis
  * active tuberculosis
  * refractory heart failure
  * previous transplantation
  * immunosuppressive therapy
  * pregnancy
  * patients with chronic pancreatitis or pancreas carcinoma
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Comparison of various scores in predicting severity and outcome in patients with acute pancreatitis. 1.Homeostatic model assessment of insulin resistance. 2.The harmless acute pancreatitis score. | within 18 months
  1. Homeostatic model assessment of insulin resistance it measure severity of insulin resistance, there is an association between insulin resistance and severity of acute pancreatitis.
     It is defined as fasting glucose (mmol/L) × fasting insulin (μmol/L)/22.5] or [fasting glucose (mg/dL) × fasting insulin (μmol/L) Reference index levels is ≤ 2. If index ˃ 2 indicate presence of insulin resistance
  2. The harmless acute pancreatitis score Harmless acute pancreatitis score contains three parameters - blood urea nitrogen, levels of serum creatinine and haematocrit . The patient is classified as harmless acute pancreatitis score negative (-) if they have blood urea nitrogen <25 mg/dL, serum creatinine levels < 2 mg/dL, and haematocrit levels of <43% for males and <39.6% for females at the time of admission. The patient is considered positive (+) if any one of the above parameters is positive.

IPD SHARING:
Plan to Share IPD: Undecided